CLINICAL TRIAL: NCT00202072
Title: Mucin in Sputum of CF During Pulmonary Exacerbation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Philipps University Marburg (Other)
Other Study IDs: 208/03
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Cystic Fibrosis
Keywords: lung; airway; pulmonary exacerbation; mucus
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to determine whether mucin is increased during pulmonay exacerbations in adult patients with cystic fibrosis (CF).

DETAILED DESCRIPTION:
CF is typically associated with mucus hypersecretion in the airways. In health, mucin is the major macromolecular component and is responsible for the protective and clearance properties of the mucus gel. In a recent study we found that mucins are decreased in the sputum of adult CF patients.

In this study we want to investigate the differences on the mucin and DNA quantity and quality of airway secretions in during pulmoanry exacerbation.We hypothesize that during an exacerbation the mucin and DNA amount is increasing.

The aim of this study is to evaluate the molecular (mucins) and structure properties (mucin-DNA-network) of the airway secretions in CF related to the severity of the disease.

We characterize sputum composition of patients with pulmonary exacerbations. Using gel electrophoresis and dot-blot with specific antibodies we will analyze MUC5AC and MUC5B mucins. DNA amount will be measured by microfluorimetry. With the laser scanning confocal microscopy the mucin-DNA-network will be evaluated.

The significance of these studies is that they will give us novel information about the pathogenesis of chronic inflammatory airway diseases, provide tools for assessing the progression of lung disease, and most critically, will identify novel opportunities and targets for therapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

* cystic fibrosis
* chronic pseudomonas aeruginosa inflammation
* pulmonary exacerbation

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2004-01; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Markus O Henke, MD, Principal Investigator — Philipps University Marburg
Locations (2):
- Germany (2):
  - Pediatric department, CF center, University Giessen, Giessen
  - Pediatric department, CF center, University Marburg, Marburg

REFERENCES:
- [Background] Henke MO, Renner A, Huber RM, Seeds MC, Rubin BK. MUC5AC and MUC5B Mucins Are Decreased in Cystic Fibrosis Airway Secretions. Am J Respir Cell Mol Biol. 2004 Jul;31(1):86-91. doi: 10.1165/rcmb.2003-0345OC. Epub 2004 Feb 26. PMID 14988081